CLINICAL TRIAL: NCT00320086
Title: Microalbuminuria in Children With and Without Diabetes
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: HRRC#04-250; M01RR000997 (NIH)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetes group: 6 to 18 years old males and females, with confirmed diagnosis of Type I or Type II Diabetes with no history of: kidney disease, documented urinary tract infection, cardiovascular disease, liver disease, nocturnal enuresis, metabolic disease other that diabetes, abnormal body temperature at start of study visit, no strenuous exercise 24 hours prior to start of study visit.
- control group: 6 to 18 years old males and females, with no history of: Type I or Type II Diabetes and/or other metabolic disease, kidney disease, documented urinary tract infection, cardiovascular disease, liver disease, nocturnal enuresis, abnormal body temperature at start of study visit, no strenuous exercise 24 hours prior to start of study visit.

SUMMARY:
The purpose of the study is to learn more about Microalbuminuria in children with and without diabetes. Albumin is a protein that may be excreted in the urine. In some conditions, like kidney problems or diabetes, the amount of albumin in the urine increases. The purpose of this study is to measure concentration of albumin in the urine of diabetic children and compare to healthy children.

DETAILED DESCRIPTION:
Diabetic nephropathy is a known cause of significant morbidity and mortality in adult patients with diabetes. Microalbuminuria (MA) is predictive of future diabetic nephropathy (DN) in adult patients with diabetes mellitus (DM). This link between MA levels and DN allows patients to receive timely interventions. The predictive value of MA for DN in children with DM, however, is not well established. Most studies looking at this association in children have only been forced to use adult MA values. Children, particularly adolescents, are known to have different normal values for 24-hour total protein excretion compared to adults and it may be that they also have different normal levels of MA. Little literature exists on normal levels of 24 hr MA in healthy children and in children with diabetes.

In this study, we seek to define the range of MA levels that falls between the 2.5 and 97.5 percentiles for children with and without DM. Once these values are established, we will have a foundation for further studies to define which, if any, MA values are predictive of DN in children. If we can establish a MA level which is predictive of DN in children, it will allow physicians to direct medical intervention at those most likely to benefit while protecting others from unnecessary medications, procedures, and risks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 6 to 18
* Diabetic children 6 to 18

Exclusion Criteria:

* kidney disease
* abnormal body temperature
* history of documented urinary tract infection
* metabolic disease other than diabetes mellitus
* circulatory disease
* liver disease
* strenuous exercise in prior 24 hours
* nocturnal enuresis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary care/specialty clinincs and community
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Jacobs, Principal Investigator — University of New Mexico- Pediatric department
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the University of New Mexico and via advertising and referral by other physicians.
Groups:
- Arm 1: Control Arm: Evaluate Normal Urinary Protein Excretion in Healthy and Diabetic Children
- Arm 2: Diabetes Arm: Children 6 to 18 years old with Type I or Type II Diabetes
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 91 | 112
Completed | 91 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Control Arm: children 6 to 18 years old without:
  * kidney disease
  * abnormal body temperature
  * history of documented urinary tract infection
  * metabolic disease
  * circulatory disease
  * liver disease
  * strenuous exercise in prior 24 hours
  * nocturnal enuresis
- Arm 2: Diabetes Arm: children 6 to 18 years old with Type I or Type II Diabetes without:
  * kidney disease
  * abnormal body temperature
  * history of documented urinary tract infection
  * metabolic disease other than diabetes mellitus
  * circulatory disease
  * liver disease
  * strenuous exercise in prior 24 hours
  * nocturnal enuresis
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 91 | 112 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91 | 112 | 203
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 57 | 102
  Male | 46 | 55 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Normal Urinary Protein Excretion in Healthy and Diabetic Children, Assessed Over 1 Day.
Time Frame: during hospitalization
Measure: Number; unit: participants
Groups:
- Arm 1: Control Arm
- Arm 2: Diabetes Arm
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 91 | 112
participants | 91 | 112
Statistical Analysis 1: Comparison: Arm 1; ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: AE data collected from study initiation to study closure. Individual Study visits: Adverse Event data was collected up to 72 hours after end of study visit. Study lab results reviewed by a study investigator as soon as received from lab.
Groups:
- Group 1: dibetes vs Healthy
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/203
Other Adverse Events (participants affected / at risk) | 0/203

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No